CLINICAL TRIAL: NCT05387369
Title: A Real World Study of Paxlovid for the Treatment of Hospitalized Patients Confirmed With COVID-19
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, Professor, Huashan Hospital
Other Study IDs: KY2022-552
Record Dates: First submitted 2022-05-23; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: paxlovid
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paxlovid: Patients with COVID-19 who visit Huashan Hospital,Fudan University from 2022 to 2027 and receive Paxlovid therapy
  Interventions: Drug: Paxlovid
- Routine therapy: Patients with COVID-19 who visit Huashan Hospital,Fudan University from 2022 to 2027 and receive routine therapy without paxlovid

INTERVENTIONS:
Drug: Paxlovid — The study is a real-world study. According to the actual medical history of patients, the usage of paxlovid will be collected.
  Groups: Paxlovid

SUMMARY:
The study was designed to analyze the efficacy and safety of Paxlovid for the treatment of COVID-19.

DETAILED DESCRIPTION:
The study is a real-world study and the case records of patients with COVID-19 who visit Huashan Hospital affiliated to Fudan University from 2022 to 2027 and receive Paxlovid therapy will be collected in this study. The medical data including patient demographic, clinical characteristics, laboratory examination, history of treatments, adverse reactions and treatment outcome will be extracted to analyze the effectivity and safety of paxlovid and explore the prognosis-relevant factors of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a positive SARS-CoV-2 test result;
* Participants who have one or more mild or moderate COVID-19 symptoms.

Exclusion Criteria:

* No specific exclusion criteria in this real world study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COVID-19 who were admitted to Huashan Hospital, Fudan University from 2022 to 2027
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Viral shedding time | up to 28 days
  time from the first positive testing to the first day of nucleic acid Ct value> 35 for both ORF1ab and N gene (in two consecutive).
Percentage of the participants who have progression of COVID-19 | up to 28 days
  Percentage of participants who experience these events by Day 28 Progress to severe and/or critical COVID-19; Death from any cause

SECONDARY OUTCOMES:
AEs and SAEs through Day 28 | up to 28 days
  Adverse events and Serious adverse events through Day 28
Percentage of participants who turned negative for SARS-CoV-2 | up to 28 days
  Percentage of participants who turned negative for SARS-COV-2 at Day 3, 5, 7, 10, 14
Time to sustained clinical recovery | up to 28 days
  Time to sustained clinical recovery

CONTACTS AND LOCATIONS:
Overall Officials: Feng Sun, MD, Principal Investigator — Huashan Hospital affliatied to Fudan University
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No